CLINICAL TRIAL: NCT06830980
Title: TMS (Transcranial Magnetic Stimulation) for Methamphetamine Use Disorder in People Living With HIV
Brief Title: Transcranial Magnetic Stimulation for Methamphetamine Use Disorder in PLWH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100353; UL1TR001998 (NIH)
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Methamphetamine Use Disorders; HIV

STUDY DESIGN:
Intervention Model Description: Within participant design with a randomized sequence of interventions.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1 (Other): Group 1 will receive actual TMS (iTBS and cTBS) on days 2 and 3 and sham TMS on day 4.
  Interventions: Device: intermittent theta burst stimulation (iTBS); Device: continuous theta burst stimulation (cTBS); Device: Sham TMS
- Group 2 (Other): Group 2 will receive actual TMS (iTBS and cTBS) on days 2 and 4 and sham TMS on day 3.
  Interventions: Device: intermittent theta burst stimulation (iTBS); Device: continuous theta burst stimulation (cTBS); Device: Sham TMS
- Group 3 (Other): Group 3 will receive sham TMS on day 2 and actual TMS (iTBS and cTBS) on days 3 and 4.
  Interventions: Device: intermittent theta burst stimulation (iTBS); Device: continuous theta burst stimulation (cTBS); Device: Sham TMS

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) — iTBS is an excitatory TMS paradigm that delivers 1800 pulses to the left dlPFC. Participants will receive 2 iTBS sessions separated by 50 minutes.
Device: continuous theta burst stimulation (cTBS) — cTBS is an inhibitory TMS paradigm that delivers 1800 pulses to the frontal pole. Participants will receive 2 iTBS sessions separated by 50 minutes.
Device: Sham TMS — Sham TMS delivered with the MagVenture B65 A/P coil

SUMMARY:
The purpose of this study is to learn more about how accelerated theta burst stimulation affects methamphetamine craving and brain activity. Theta burst stimulation is a unique transcranial magnetic stimulation (TMS) paradigm that is efficient and potent.

DETAILED DESCRIPTION:
The investigators will compare how two theta burst paradigms, intermittent theta burst stimulation (iTBS) and continuous theta burst stimulation (cTBS), compare with sham TMS in changing methamphetamine craving and brain activity. iTBS, cTBS, and sham TMS will be delivered in an accelerated fashion (two sessions daily, separated by 50 minutes). iTBS will be delivered to the left dorsolateral prefrontal cortex (left dorsolateral prefrontal cortex), and cTBS will be delivered to the frontal pole. A brain MRI scan will be done before and after the iTBS/cTBS/sham TMS sessions. The study involves four visits. Each visit will last three hours. Hence, participants will spend a total of 12 hours in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults in the age group 18-65 years
* Able to read and understand English
* Able to provide informed consent
* Diagnosed with HIV
* History of current or previous Methamphetamine Use Disorder
* Endorse craving for methamphetamine
* Demonstrate an attentional bias for methamphetamine

Exclusion Criteria:

* Traumatic brain injury
* h/o seizure disorder
* h/o or current diagnosis of schizophrenia
* intracranial metal shrapnel
* previous adverse effects with TMS
* sub-threshold consistency while performing behavioral tasks
* lack of attentional bias to methamphetamine cues
* a positive pregnancy test for female participants
* abnormal brain MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cue-induced methamphetamine craving | Baseline and before and after each TMS session up to 4 days
  Measured on the visual analog scale (VAS) Scored 0 to 100 with 0=no craving and 100=the most craving.

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, MD, Principal Investigator — University of Kentucky
Locations (1):
- UK Department of Psychiatry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao D, Li Y, Liu T, Voon V, Yuan TF. Twice-Daily Theta Burst Stimulation of the Dorsolateral Prefrontal Cortex Reduces Methamphetamine Craving: A Pilot Study. Front Neurosci. 2020 Mar 25;14:208. doi: 10.3389/fnins.2020.00208. eCollection 2020. PMID 32273837
- [Background] Wen Y, Li Y, Jiang F, Dong X. TBS combined with virtual-reality reconsolidation intervention for methamphetamine use disorder: A pilot study. Brain Stimul. 2022 Jul-Aug;15(4):996-998. doi: 10.1016/j.brs.2022.07.001. Epub 2022 Jul 12. No abstract available. PMID 35835436
- [Background] Wang W, Zhu Y, Wang L, Mu L, Zhu L, Ding D, Ren Z, Yang D, Tang H, Zhang L, Song P, Wei H, Chang L, Wang Z, Ling Q, Gao H, Liu L, Jiao D, Xu H. High-frequency repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex reduces drug craving and improves decision-making ability in methamphetamine use disorder. Psychiatry Res. 2022 Nov;317:114904. doi: 10.1016/j.psychres.2022.114904. Epub 2022 Oct 12. PMID 36265196
- [Background] van Rooij SJH, Arulpragasam AR, McDonald WM, Philip NS. Accelerated TMS - moving quickly into the future of depression treatment. Neuropsychopharmacology. 2024 Jan;49(1):128-137. doi: 10.1038/s41386-023-01599-z. Epub 2023 May 22. PMID 37217771
- [Background] Suppa A, Huang YZ, Funke K, Ridding MC, Cheeran B, Di Lazzaro V, Ziemann U, Rothwell JC. Ten Years of Theta Burst Stimulation in Humans: Established Knowledge, Unknowns and Prospects. Brain Stimul. 2016 May-Jun;9(3):323-335. doi: 10.1016/j.brs.2016.01.006. Epub 2016 Jan 27. PMID 26947241
- [Background] Su H, Chen T, Jiang H, Zhong N, Du J, Xiao K, Xu D, Song W, Zhao M. Intermittent theta burst transcranial magnetic stimulation for methamphetamine addiction: A randomized clinical trial. Eur Neuropsychopharmacol. 2020 Feb;31:158-161. doi: 10.1016/j.euroneuro.2019.12.114. Epub 2020 Jan 2. PMID 31902567
- [Background] Rakesh G, Adams TG, Morey RA, Alcorn JL 3rd, Khanal R, Su AE, Himelhoch SS, Rush CR. Intermittent theta burst stimulation and functional connectivity in people living with HIV/AIDS who smoke tobacco cigarettes: a preliminary pilot study. Front Psychiatry. 2024 Mar 4;15:1315854. doi: 10.3389/fpsyt.2024.1315854. eCollection 2024. PMID 38501083
- [Background] Mehta DD, Praecht A, Ward HB, Sanches M, Sorkhou M, Tang VM, Steele VR, Hanlon CA, George TP. A systematic review and meta-analysis of neuromodulation therapies for substance use disorders. Neuropsychopharmacology. 2024 Mar;49(4):649-680. doi: 10.1038/s41386-023-01776-0. Epub 2023 Dec 12. PMID 38086901
- [Background] Liu Q, Sun H, Hu Y, Wang Q, Zhao Z, Dong D, Shen Y. Intermittent Theta Burst Stimulation vs. High-Frequency Repetitive Transcranial Magnetic Stimulation in the Treatment of Methamphetamine Patients. Front Psychiatry. 2022 Apr 26;13:842947. doi: 10.3389/fpsyt.2022.842947. eCollection 2022. PMID 35558419
- [Background] Geoly AD, Kratter IH, Toosi P, Cole EJ, Sahlem GL, Williams NR. Sustained Efficacy of Stanford Neuromodulation Therapy (SNT) in Open-Label Repeated Treatment. Am J Psychiatry. 2024 Jan 1;181(1):71-73. doi: 10.1176/appi.ajp.20230113. No abstract available. PMID 38161297
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Chen T, Su H, Wang L, Li X, Wu Q, Zhong N, Du J, Meng Y, Duan C, Zhang C, Shi W, Xu D, Song W, Zhao M, Jiang H. Modulation of Methamphetamine-Related Attention Bias by Intermittent Theta-Burst Stimulation on Left Dorsolateral Prefrontal Cortex. Front Cell Dev Biol. 2021 Aug 3;9:667476. doi: 10.3389/fcell.2021.667476. eCollection 2021. PMID 34414178
- [Background] Chen T, Su H, Li R, Jiang H, Li X, Wu Q, Tan H, Zhang J, Zhong N, Du J, Gu H, Zhao M. The exploration of optimized protocol for repetitive transcranial magnetic stimulation in the treatment of methamphetamine use disorder: A randomized sham-controlled study. EBioMedicine. 2020 Oct;60:103027. doi: 10.1016/j.ebiom.2020.103027. Epub 2020 Sep 25. PMID 32980696
- [Background] Ballester J, Marchand WR, Philip NS. Transcranial magnetic stimulation for methamphetamine use disorder: A scoping review within the neurocircuitry model of addiction. Psychiatry Res. 2024 Aug;338:115995. doi: 10.1016/j.psychres.2024.115995. Epub 2024 May 29. PMID 38852478